CLINICAL TRIAL: NCT00679835
Title: An Evaluation of the Pharmacokinetic Profile and Safety of a Single Dose of Daptomycin in Pediatric Subjects Aged Two to Six Years Who Are Concurrently Receiving Standard Antibiotic Therapy for Proven or Suspected Gram-positive Infection
Brief Title: PK and Safety Evaluation of Daptomycin in Children Ages 2-6 With Proven or Suspected Gram-positive Infections
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 3009-023; DAP-PEDS-07-02 (Other: Cubist Study Number)
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Gram Positive Infection; Concurrent Antibiotic Treatment
MeSH Terms: interventions — Daptomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): 8 mg/kg over a one hour infusion
  Interventions: Drug: daptomycin
- Group 2 (Experimental): 10mg/kg over a one or two hour infusion
  Interventions: Drug: daptomycin

INTERVENTIONS:
Drug: daptomycin — i.v. daptomycin given at 8 mg/kg or 10 mg/kg by a one or two hour infusion.
  Other Names: Cubicin

SUMMARY:
This is a research study designed to look at the pharmacokinetics (distribution, breakdown, and removal) and tolerability of a single dose of daptomycin in patients aged 2 to 6 years who have infections that are caused by a specific group of bacteria (called Gram-positive bacteria).

ELIGIBILITY:
Inclusion Criteria:

* Written parental (or appropriate legal representative) informed consent prior to any study-related procedure not part of normal medical care;
* Male or female between the ages of 2 and 6 years old, inclusive;
* Able to comply with the protocol for the duration of the study;
* Clinically stable with no evidence of hemodynamic instability (defined as a requirement for pharmacological intervention to manage blood pressure) in the 72 hour window prior to enrollment, and no history or evidence of renal or hepatic compromise;
* Suspected or diagnosed Gram-positive infection for which the subject is receiving standard antibiotic therapy;
* A calculated creatinine clearance rate (CLcr) ≥ 80 ml/min/1.73m2 as determined by the Schwartz equation at baseline;
* Creatine phosphokinase (CPK) levels less than 2X ULN (upper limit of normal) at baseline.
* Presence of two patent intravenous lines (or comparable means of venous access) prior to dosing on Study Day 1.

Exclusion Criteria:

* Investigational drug use (including daptomycin) or participation in any experimental procedure in the 30 days preceding study entry;
* Known allergy/ hypersensitivity to daptomycin;
* History of clinically significant cardiovascular, renal, hepatic, pulmonary (well-controlled asthma is acceptable), gastrointestinal, endocrine, hematologic, autoimmune disease or primary immune deficiency;
* Pneumonia as sole Gram-positive infection being treated with standard antibiotics;
* Subjects with clinically significant abnormal laboratory test results [including electrocardiograms (ECGs)], as determined by Investigator;
* Administration of rifampin within 7 days of study drug administration;
* Body mass index (BMI) that is outside of the 5th to 95th percentile;
* Subjects in whom collection of the required blood volume would put them at risk of hemodynamic disturbance (at the discretion of Investigator);
* History of or current clinically significant (at the discretion of the Investigator) muscular disease, nervous system or seizure disorder;
* Administration of intramuscular injection between baseline and study drug administration or expected intramuscular injection within 24 hours following dosing;
* Expected surgical procedure(s) within 24 hours prior to and following dosing;
* Unexplained muscular weakness, history of peripheral neuropathy, Guillian-Barre or spinal cord injury;
* History of or current rhabdomyolysis.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2008-06-03 (Actual); Primary Completion 2008-11-20 (Actual); Study Completion 2008-11-20 (Actual)

PRIMARY OUTCOMES:
Pharmocokinetics of daptomycin | From pre-dose to 24 hours post-dose

SECONDARY OUTCOMES:
Safety of daptomycin | Up to 9 days after dosing

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Abdel-Rahman SM, Chandorkar G, Akins RL, Bradley JS, Jacobs RF, Donovan J, Benziger DP. Single-dose pharmacokinetics and tolerability of daptomycin 8 to 10 mg/kg in children aged 2 to 6 years with suspected or proved Gram-positive infections. Pediatr Infect Dis J. 2011 Aug;30(8):712-4. doi: 10.1097/INF.0b013e31820fc8e1. PMID 21317681